CLINICAL TRIAL: NCT04899115
Title: A Randomized Controlled Trial of VE303 to Treat Hepatic Encephalopathy
Brief Title: VE303 for Treatment of Hepatic Encephalopathy (HE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patricia Bloom (Other)
Collaborators: Vedanta Biosciences, Inc. (Industry); American College of Gastroenterology (Other); American Association for the Study of Liver Diseases (Other)
Responsible Party: Sponsor-Investigator, Patricia Bloom, Clinical Lecturer in Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00194437
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy | interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 to VE303 vs placebo. There will be no stratification.
  After the trial enrolls the first 9 patients, an interim analysis to evaluate safety of VE303 in this population will take place. If there is no concern for a higher rate of Serious adverse events (SAEs) in the VE303 group, enrollment will continue to reach a total of 18 patients.
Who Masked: Participant, Investigator
Masking Description: Study staff will remain blinded to subject randomization until the study period is over.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: oral vancomycin
- VE303 (Experimental): VE303 is a live biotherapeutic product comprising 8 nonpathogenic commensal strains of Clostridia.
  Interventions: Drug: VE303; Drug: oral vancomycin

INTERVENTIONS:
Drug: Placebo — Starting the last day of oral vancomycin (Day 1), subjects randomized to this arm will take 5 capsules of placebo for 14 days taken once daily.
  Arms: Placebo
Drug: VE303 — Starting the last day of oral vancomycin (Day 1), subjects randomized to this arm will take 5 capsules of VE303 taken daily for 14 days.
  The quantity of each strain is proportioned to assure a specific per-strain per-capsule titer. The 8 strains are blended together with a micro-crystalline cellulose flow agent and placed in enteric capsules.
  Arms: VE303
Drug: oral vancomycin — All enrolled subjects will receive 5 days of oral vancomycin 125 mg four times a day (q.i.d).

SUMMARY:
This research is studying the use of a new drug to learn about its safety and efficacy as a treatment for hepatic encephalopathy.

Eligible participants will be enrolled and given oral antibiotics followed by 14 days of the study drug (placebo vs.VE303). There will be visits as well as other procedures to collect blood and stool samples, and have tests of your cognition (thinking) for this research study.

The hypothesis is that VE303 will safely and effectively improve cognitive function in patients with a history of overt hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cirrhosis based on liver biopsy, imaging, or evidence of clinical decompensation
* History of at least one episode of overt HE any time in the past
* Prescribed both lactulose and rifaximin, and compliant with this treatment

Exclusion Criteria:

* Current episode of overt HE
* Variceal bleeding in the last 4 weeks
* Gut-absorbable or intravenous antibiotic therapy in the last 28 days
* Fecal microbiota transplant in the last 6 months
* Use of probiotics in the last 2 weeks
* Alcohol or illicit drug intake in the last 4 weeks
* Primary sclerosing cholangitis as etiology of liver disease
* History of inflammatory bowel disease, short gut, gastrointestinal tract fistulas, intestinal ischemia, or any form of ongoing colitis
* Prior diagnosis of dementia or other primary neurocognitive disorder
* Known hypersensitivity/allergy/intolerance to Vancomycin and any ingredients of VE303: sucrose, histidine, yeast extract, cysteine, metabisulfite, and microcrystalline cellulose
* History of Roux-en-Y Gastric bypass
* Any gastrointestinal surgery in the last year
* Substantial immune compromise/deficiency (e.g., uncontrolled human immunodeficiency virus, active immune suppressive therapy including high doses of corticosteroids or medications to prevent graft rejection, recent myeloablative therapy, sustained neutropenia)
* Pregnancy or breast feeding
* Model for end-stage liver disease (MELD) > 20
* History of spontaneous bacterial peritonitis
* Hemodialysis in the last 28 days
* Placement of a portosystemic shunt or transjugular intrahepatic portosystemic shunt in the last 3 months (permissible if placed >3 months before enrollment)
* Unstable doses of opiates, benzodiazepines or other sedating medication
* Chronic methadone or low dose benzodiazepines (for example) is acceptable

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bloom, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was consented but then failed to meet eligibility criteria soon after enrollment. They did not initiate vancomycin and were not randomized.
Groups:
- Placebo: Placebo: Starting the last day of oral vancomycin (Day 1), participants randomized to this arm will take 5 capsules of placebo for 14 days taken once daily.
  Oral vancomycin: All enrolled participants will receive 5 days of oral vancomycin 125 mg four times a day (q.i.d).
- VE303: VE303 is a live biotherapeutic product comprising 8 nonpathogenic commensal strains of Clostridia.
  VE303: Starting the last day of oral vancomycin (Day 1), participants randomized to this arm will take 5 capsules of VE303 taken daily for 14 days.
  The quantity of each strain is proportioned to assure a specific per-strain per-capsule titer. The 8 strains are blended together with a micro-crystalline cellulose flow agent and placed in enteric capsules.
  Oral vancomycin: All enrolled subjects will receive 5 days of oral vancomycin 125 mg four times a day (q.i.d).
Period: Overall Study
Arm/Group | Placebo | VE303
Started | 6 | 12
Completed | 6 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VE303: VE303 is a live biotherapeutic product comprising 8 nonpathogenic commensal strains of Clostridia.
  VE303: Starting the last day of oral vancomycin (Day 1), participants randomized to this arm will take 5 capsules of VE303 taken daily for 14 days.
  The quantity of each strain is proportioned to assure a specific per-strain per-capsule titer. The 8 strains are blended together with a micro-crystalline cellulose flow agent and placed in enteric capsules.
  Oral vancomycin: All enrolled participants will receive 5 days of oral vancomycin 125 mg four times a day (q.i.d).
- Total: Total of all reporting groups
Arm/Group | Placebo | VE303 | Total
Number analyzed (Participants) | 6 | 12 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (7) | 58 (10) | 60 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 4 | 6 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 2
  White | 4 | 10 | 14
  Other | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 12 | 18
Baseline Psychometric HE Score (PHES) [Mean (Standard Deviation); unit: units on a scale] — This score is a battery of 5 paper-pencil tests that evaluate cognitive and psychomotor processing speed and visuomotor coordination. Scores on each subtest are assigned values based on age-related norms (1+ for scores better than 1 standard deviation (SD) above the normal mean to -3 for scores more than 3 SDs below the normal mean). Combined scores vary from +6 to -18, where +6 is the best function and -18 is worst function
  units on a scale | -5.0 (3.7) | -6.3 (3.4) | -5.8 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Serious Adverse Events up to Week 6
Description: An adverse event (AE) or suspected adverse reaction is considered "serious" if, in the view of the investigator, it results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Week 6
Measure: Count of Participants; unit: Participants
Arm/Group | VE303 | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 2 | 0

2. Primary Outcome: Change in Psychometric Hepatic Encephalopathy Score (PHES) as a Measure of Cognitive Function From Pre-vancomycin to Week 6
Description: This score is a battery of 5 paper-pencil tests that evaluate cognitive and psychomotor processing speed and visuomotor coordination. Scores on each subtest are assigned values based on age-related norms (1+ for scores better than 1 standard deviation (SD) above the normal mean to -3 for scores more than 3 SDs below the normal mean). Combined scores vary from +6 to -18, where +6 is the best function and -18 is worst function.
Time Frame: baseline (pre-vancomycin), Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- VE303: VE303 is a live biotherapeutic product comprising 8 nonpathogenic commensal strains of Clostridia.
  VE303: Starting the last day of oral vancomycin (Day 1), subjects randomized to this arm will take 5 capsules of VE303 taken daily for 14 days.
  The quantity of each strain is proportioned to assure a specific per-strain per-capsule titer. The 8 strains are blended together with a micro-crystalline cellulose flow agent and placed in enteric capsules.
  oral vancomycin: All enrolled subjects will receive 5 days of oral vancomycin 125 mg four times a day (q.i.d).
Arm/Group | Placebo | VE303
Number analyzed (Participants) | 6 | 12
units on a scale | -1.0 (3.7) | 1.5 (3.5)

3. Secondary Outcome: Number of Hospitalizations for Overt Hepatic Encephalopathy (OHE) up to Week 26
Description: Shown as a rate (# of episodes/ number of patients) = # per patient.
Time Frame: 26 weeks
Measure: Mean (Full Range); unit: episodes/patient
Arm/Group | Placebo | VE303
Number analyzed (Participants) | 6 | 12
episodes/patient | .333 [0 to 2] | 1.25 [0 to 6]

4. Secondary Outcome: Adverse Events up to Week 26
Description: total number of AEs
Time Frame: up to week 26
Measure: Number; unit: adverse events
Arm/Group | Placebo | VE303
Number analyzed (Participants) | 6 | 12
adverse events | 38 | 135

5. Secondary Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS) Global Health Reported From Pre-vancomycin to Week 26
Description: The PROMIS v 1.1 is a 10 question scale where participants select answers from (0) up to (10). Higher scores indicate better quality of life. Results are presented as change in scores pertaining to physical and mental health.
Time Frame: baseline (pre-vancomycin), week 26
Population: Data is missing from two VE303 participants because they did not provide it.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | VE303
Number analyzed (Participants) | 6 | 10
score on a scale
  Change in PROMIS Physical Health Scores | 1.8 (1.8) | 0.4 (1.9)
  Change in PROMIS Mental Health Scores | 1.2 (2.1) | 0 (2.4)

6. Secondary Outcome: Time to Overt HE
Description: This is the number of days from Day 1 of Vancomycin to the first OHE event or to the end of study, whichever came first.
Time Frame: up to 26 weeks
Measure: Mean (Full Range); unit: days
Arm/Group | Placebo | VE303
Number analyzed (Participants) | 6 | 12
days | 180 [170 to 182] | 147 [16 to 182]

7. Secondary Outcome: Change in Microbiome Composition From Pre-vancomycin to Week 26
Description: This will be calculated by alpha diversity between stool collection timepoints and will have metagenomic sequencing on stool to assess this. The Shannon index is a calculation used to measure the diversity of microbial species within a sample, taking into account both the number of different species present (richness) and how evenly distributed their abundances are (evenness). A higher Shannon index indicates a more diverse microbial community, meaning a wider variety of microbes present in roughly equal proportions. The Shannon index was calculated for each sample as part of metagenomic sequencing analysis performed with the tool MetaPhlAn (version 3.0). The minimum Shannon index value is 0 and it could theoretically go to infinity; however, typical values range more in the 1-4 range. Now, this outcome is measuring the CHANGE in Shannon index, therefore negative values are possible, if the diversity of specimens dropped from the pre-vancomycin to the week 26 samples.
Time Frame: baseline (pre-vancomycin), week 26
Population: Participants analyzed reflect participants from whom week 26 stool samples could be obtained. Not every participant was able to provide a stool sample at week 26, and therefore this outcome was missing for those patients.
Measure: Mean (Standard Deviation); unit: Shannon index
Arm/Group | VE303 | Placebo
Number analyzed (Participants) | 6 | 2
Shannon index | 0.37 (0.72) | -0.15 (0.06)
Statistical Analysis 1: Comparison: VE303 vs Placebo; Test type: Superiority; p = 0.13, t-test, 2 sided

8. Secondary Outcome: PHES From Pre-vancomycin to Week 26
Description: This score is a battery of 5 paper-pencil tests that evaluate cognitive and psychomotor processing speed and visuomotor coordination. Scores on each subtest are assigned values based on age-related norms (+1 for scores better than 1 standard deviation (SD) above the normal mean to -3 for scores more than 3 SDs below the normal mean). Combined scores vary from +6 to -18.
Time Frame: pre-vancomycin up to week 26
Population: Note: Significant data loss due to some participants not participating in this test at 26 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Placebo | VE303
Number analyzed (Participants) | 4 | 9
score on a scale | -1 [-3 to 1] | 1 [-6 to 10]
Statistical Analysis 1: Comparison: Placebo vs VE303; Test type: Superiority; p = 0.48, Wilcoxon (Mann-Whitney); Wilcoxon was used because data was not normal

9. Other Pre Specified Outcome: Change in Serum and Stool Biomarkers From Pre-vancomycin to Week 26
Time Frame: baseline (pre-vancomycin), week 26
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Placebo | VE303
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/6 | 5/12
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | VE303 (N=12)
Hospitalized for Hepatic Encephalopathy (Hepatobiliary disorders) | 1 | 4
Inpatient Catheter Service (Surgical and medical procedures) | 0 | 1
Hyperglycemic Hyperosmolar Syndrome (Metabolism and nutrition disorders) | 0 | 1
Hospitalization due to Ascites Accumulation (Hepatobiliary disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Hospitalization for Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 — This adverse event occurred in conjunction with others
Pain and Bleeding from Surgical Site (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Hospitalization due to Esophageal Bleed (Gastrointestinal disorders) | 1 | 0
Elective Total Hip Replacement (Surgical and medical procedures) | 0 | 1
Hospitalization due to Post-Surgical Complications (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | VE303 (N=12)
Abdominal Distension (Gastrointestinal disorders) | 0 | 7 — This adverse event occurred in conjunction with others
Increased Bowel Movements (Gastrointestinal disorders) | 1 | 5
Bradycardia (Cardiac disorders) | 0 | 1
Bruising (Skin and subcutaneous tissue disorders) | 0 | 3
Fatigue (General disorders) | 1 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 7 — This adverse event occurred in conjunction with others
Decreased Lymphocyte Count (Blood and lymphatic system disorders) | 1 | 7
Decreased Platelet Count (Blood and lymphatic system disorders) | 3 | 3
Alkaline Phosphatase Increase (Hepatobiliary disorders) | 2 | 3
Worsening Gout Symptoms (Musculoskeletal and connective tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 8 — This adverse event occurred in conjunction with others
Alanine Transaminase Increase (Hepatobiliary disorders) | 2 | 0
Increased Blood Bilirubin (Hepatobiliary disorders) | 1 | 3
Increased Lipase (Gastrointestinal disorders) | 2 | 4
Leukopenia/Decreased White Blood Cell Count (Blood and lymphatic system disorders) | 1 | 3
Chills (General disorders) | 0 | 3 — This adverse event occurred in conjunction with others
Nausea (Gastrointestinal disorders) | 1 | 7 — This adverse event occurred in conjunction with others
Increased Amylase Levels (Gastrointestinal disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Skin Numbness (Skin and subcutaneous tissue disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 3
Hypokalemia (Metabolism and nutrition disorders) | 0 | 4
Leg Pain and Swelling (General disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Skin Discoloration (foot) (Skin and subcutaneous tissue disorders) | 0 | 1
Easy Bleeding (Blood and lymphatic system disorders) | 0 | 1
Long Sleeping Duration (General disorders) | 1 | 0
Limb Weakness/Numbness (Nervous system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 3
Decreased Neutrophil Count (Blood and lymphatic system disorders) | 1 | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 | 1
Bilateral Hand Tremors (Nervous system disorders) | 0 | 1 — This adverse event occurred in conjunction with others
Flatulence (Gastrointestinal disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Lightheadedness (General disorders) | 0 | 1 — This adverse event occurred in conjunction with others
Weight Gain (General disorders) | 0 | 1
Flu Symptoms (Infections and infestations) | 0 | 1
Mild Edema (General disorders) | 0 | 1
COVID (Infections and infestations) | 0 | 1 — This adverse event occurred in conjunction with others
Bleeding from preexisting ear condition (Ear and labyrinth disorders) | 1 | 0
Eosinophilia (Immune system disorders) | 1 | 1
Ear Ache post Ear AVM ablation (Ear and labyrinth disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hot Flashes/Night Sweats (General disorders) | 0 | 2
Increased INR (Blood and lymphatic system disorders) | 0 | 2
Weight Loss (General disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3
Difficulty Falling Asleep (General disorders) | 0 | 1
Increased Creatinine (Renal and urinary disorders) | 0 | 1
Disorientation (Nervous system disorders) | 0 | 1
Slow Speech (Nervous system disorders) | 0 | 1
Asterixis (Nervous system disorders) | 0 | 1
Headache (General disorders) | 1 | 4 — This adverse event occurred in conjunction with others
Loss of Appetite (General disorders) | 1 | 0
Increase in Aspartate Aminotransferase (Hepatobiliary disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Note that for PHES and some other outcome measures, the drop out rate was high.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/15/NCT04899115/Prot_SAP_000.pdf